CLINICAL TRIAL: NCT00164866
Title: Administration of Intravenous Proton Pump Inhibitor Prior to Endoscopy [APPE] in Patients With Upper Gastrointestinal Bleeding; a Double-Blind Placebo-Controlled Randomised Study.
Brief Title: Administration of High-Dose Intravenous Proton Pump Inhibitor for Upper Gastrointestinal Bleeding Prior to Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPE
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-06

CONDITIONS: Peptic Ulcer
Keywords: Peptic ulcer; IVPPI prior endoscopy
MeSH Terms: conditions — Peptic Ulcer | interventions — Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
To evaluate if intravenous PPI infusion, when administered prior to endoscopy, hastens resolution of bleeding stigmata and thereby facilitates endoscopic examinations and reduces the need for endoscopic treatment. Clot stabilization may itself sustain control of bleeding before endoscopy. These may translate into improved patients'outcome and survival.

To determine the therapeutic effect of high-dose PPI infusion in upper gastrointestinal bleeding from causes other than peptic ulcers.

DETAILED DESCRIPTION:
A placebo-controlled randomised study is being proposed. We hypothesize that early administration of intravenous omeprazole infusion stabilizes clots overlying arteries and hastens resolution of bleeding stigmata in peptic ulcer, and facilitates subsequent endoscopic examinations and reduces the need for endoscopic treatment. This may translates into clinical benefits in those who receive early intravenous omeprazole.

Consecutive patients with overt signs of upper gastrointestinal bleeding will be randomised to receive omeprazole or its equivalent placebo (80mg i.v. bolus followed by 8mg/hr) until next scheduled endoscopy. Patients with circulatory instability or fresh hematemesis will undergo endoscopic examinations urgently after initial stabilisation. The infusion will continue until endoscopic examination with or without therapy. Next scheduled endoscopy is performed within 24 hours from admission by experienced endoscopists with expertise in therapeutic endoscopy. At endoscopy, actively bleeding ulcers or ulcers with non-bleeding visible vessels are to be treated by endoscopic therapy. Omeprazole infusion 8mg/hr is to be continued for 72 hours after endoscopic hemostasis.

Patients will be followed-up for 30 days from the time of admission or if patients stay longer than 30 days, the time to hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with overt signs of upper GIB; fresh hematemesis and/or melena with or with circulatory compromise

Exclusion Criteria:

* Chronic aspirin user,
* Pregnancy,
* Age<16,
* Allergy to PPI,
* No consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 638
Dates: Start 2004-02; Study Completion 2005-09

PRIMARY OUTCOMES:
early intranvenous infusion of a high-dose poton-pump inhibitor before endoscopy would have a therapeutic effect on bleeding ulcers, reduce the need for endoscopic therapy, and result in improved clinical outcomes.

SECONDARY OUTCOMES:
Control of bleeding (absence of active bleeding) at the time of endoscopic procedure
The prevalence of stigmata of bleeding at endoscopic examination
30-day survival
Hospital stay
Transfusion requirement

CONTACTS AND LOCATIONS:
Overall Officials: James Y Lau, MD, Principal Investigator — Endoscopy Center, Prince of Wales Hospital
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Derived] Tsoi KK, Lau JY, Sung JJ. Cost-effectiveness analysis of high-dose omeprazole infusion before endoscopy for patients with upper-GI bleeding. Gastrointest Endosc. 2008 Jun;67(7):1056-63. doi: 10.1016/j.gie.2007.11.056. Epub 2008 Apr 14. PMID 18407271
- [Derived] Lau JY, Leung WK, Wu JC, Chan FK, Wong VW, Chiu PW, Lee VW, Lee KK, Cheung FK, Siu P, Ng EK, Sung JJ. Omeprazole before endoscopy in patients with gastrointestinal bleeding. N Engl J Med. 2007 Apr 19;356(16):1631-40. doi: 10.1056/NEJMoa065703. PMID 17442905